CLINICAL TRIAL: NCT06730906
Title: Testing and Refinement of PACTAID App in Patients With Type 1 Diabetes to Help Manage Exercise While on Automated Insulin Delivery System
Brief Title: PACTAID App in Adults With Type 1 Diabetes to Help Manage Exercise
Acronym: PACTAID
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Arizona State University (Other); University of Houston (Other)
Responsible Party: Principal Investigator, Yogish C. Kudva, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 24-007866
Record Dates: First submitted 2024-12-05; First posted 2024-12-12 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: T1D; Type 1 Diabetes; Type 1 Diabetes Mellitus; Exercise; automated insulin delivery
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention Group (Experimental): Participants will utilize the PACTAID app for 8 weeks.
  Interventions: Device: PACTAID App

INTERVENTIONS:
Device: PACTAID App — The PACTAID app will provide real time decision support during exercise for patients with type 1 diabetes.

SUMMARY:
The purpose of this trial is to test and refine the PACTAID smart phone application in adults with type 1 diabetes mellitus to help manage exercise while on automated insulin delivery systems with the goal of improving glycemic control during and after exercise as well as improving multiple other cardiovascular risk factors.

DETAILED DESCRIPTION:
This trial will be conducted in two phases. In Phase 1, we will test the PACTAID app in adults with type 1 diabetes mellitus to help manage exercise while on an automated insulin delivery system for four weeks. In phase 2, we will use a refined version of the PACTAID app in those same adults from phase 1 for four weeks. A 2-4-week period will be between phase 1 and phase 2 in which the app will be refined. There is one clinical site, Mayo Clinic, and two sites creating the app, Arizona State University and University of Houston. The study will enroll up to 8 subjects at Mayo Clinic.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female between age of 18-65 yrs.
* T1D diagnosis will be confirmed by C- Peptide (≤0.6 ng/ml) with a simultaneous fasting glucose concentration 80-225 mg/dL.
* T1D using AID either tandem Control IQ, Medtronic 780G, Omnipod 5 or Ilet bionic pancreas for diabetes management at the time of screening for at least 3-month duration.
* CGM and insulin pump data available for > 70% for last 2 weeks.
* T1D without atherosclerotic cardiovascular disease
* HbA1c ≤10 %
* Able to understand English language.
* Currently using an insulin-to-carbohydrate ratio to calculate meal bolus sizes.
* Willing to complete study procedures.
* Willing to wear study devices.
* An understanding of and willingness to follow the protocol, perform all 3 types of exercises as per protocol, and sign the informed consent.
* Non-smoker
* Satisfactory EKG in last one year or if not available, satisfactory baseline EKG at screening

Exclusion Criteria:

* Anti-hyperglycemic drugs other than insulin including metformin.
* Pregnancy or contemplating pregnancy in study
* Untreated hyperthyroidism or hypothyroidism, abnormal (out of Reference range) TSH at the time of screening
* Severe hypoglycemia or DKA in last 3 months.
* Baseline exercise status-those already doing vigorous exercise such as 1 hour per day will be excluded.
* BMI ≥35 kg/m2
* Obstructive sleep apnea not controlled on CPAP.
* Chronic obstructive pulmonary disease
* Asthma limiting exercise.
* Uncontrolled hypertension, Blood pressure ≥ 140/90 mmHg with ≥ 2 antihypertensive medications
* Clinically diagnosed obstructive coronary artery disease or any other significant cardiac condition or heart failure
* Uncontrolled or recurrent ventricular tachycardia
* Any medication affecting heart rate.
* Clinical diagnosis of unstable proliferative diabetic retinopathy
* Previous Organ Transplant with or without current graft function
* Currently receiving chemotherapy or long-term immunosuppressant (glucocorticoids etc.) therapy
* COVID positive at the time of screening
* Clinically diagnosed autonomic neuropathy
* Abnormal liver function test results (Transaminase >3 times the upper limit of normal); testing required for subjects taking medications known to affect liver function or with diseases known to affect liver function.
* Abnormal renal function test results (calculated GFR <60 mL/min/1.73m2)
* Active gastroparesis
* Abuse of alcohol or recreational drugs
* Infectious process not anticipated to resolve prior to study procedures (e.g., meningitis, pneumonia, osteomyelitis).
* If on anti-depressant, lack of stability on the medication for the past 2 months prior to enrollment in the study
* Any known medical condition that in the judgment of the investigator might interfere with the completion of the protocol such as the following examples:

  1. Inpatient psychiatric treatment in the past 6 months
  2. Presence of a known adrenal disorder
  3. A recent injury to body or limb, muscular disorder, use of any medication, any carcinogenic disease, or other significant medical disorder if that injury, medication, or disease in the judgment of the investigator will affect the completion of the protocol
  4. Participating in any other treatment study

Note: Other protocol defined Inclusion/Exclusion Criteria may apply.

Eligibility last updated 08/15/2024. Questions regarding updates should be directed to the study team contact.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-01-10 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Mean CGM glucose (mg/dL) | Baseline, 4 weeks, 8 weeks
  Change in mean CGM glucose (mg/dL)
CGM glucose SD (mg/dL) | Baseline, 4 weeks, 8 weeks
  Change in CGM glucose SD (mg/dL)
Glucose coefficient of variation (%) | Baseline, 4 weeks, 8 weeks
  Change in glucose coefficient of variation (%)
CGM TIR (70-180mg/dL) | Baseline, 4 weeks, 8 weeks
  Change in CGM TIR (70-180mg/dL)
CGM TBR (<70 and <54 mg/dL) | Baseline, 4 weeks, 8 weeks
  Change in CGM TBR (<70 and <54 mg/dL)
CGM TAR (>180 and >250 mg/dL) | Baseline, 4 weeks, 8 weeks
  Change in CGM TAR (>180 and >250 mg/dL)

SECONDARY OUTCOMES:
Adherence to exercise | Baseline, 8 weeks
  Data will be collected via the PACTAID app, which will generate reports on the number of exercise sessions logged by patients. Since participants will also be wearing a Fitbit watch, we will capture heart rate changes during exercise, which will help confirm their physical activity. Furthermore, participants will complete the International Physical Activity Questionnaire (IPAQ) approximately once a month throughout the study.
CGM hypoglycemic events | Baseline, 8 weeks
  Frequency of CGM measured Hypoglycemic events
Severe hypoglycemia | Baseline, 8 weeks
  Frequency of severe hypoglycemia (requiring assistance from another person to recover from hypoglycemia)
Ambulatory blood pressure | Baseline, 8 weeks
  Change in ambulatory blood pressure
Ambulatory Arterial Stiffness Index | Baseline, 8 weeks
  Change in ambulatory arterial stiffness Index
HsCRP | Baseline, 8 weeks
  Change in HsCRP
Body weight or BMI | Baseline, 8 weeks
  Change in body weight or BMI

OTHER OUTCOMES:
App confidence | Baseline, 8 weeks
  Confidence with app use during the exercise
Fear of hypoglycemia | Baseline, 8 weeks
  The severity of hypoglycemia will be assessed monthly using the Clarke Hypoglycemia Unawareness Questionnaire. Additionally, participants will have the opportunity to add comments in the app before or after exercise sessions to indicate if they chose not to exercise due to concerns about hypoglycemia.
Step count | Baseline, 8 weeks
  Step count will be assessed by a FitBit. We will assess the correlation of step count on CGM glucose metrics (TIR, TAR and TBR)
Heart rate | Baseline, 8 weeks
  Heart rate will be assessed by a Fitbit. We will assess heart rate to determine if there is a relationship between CGM glucose metrics (TIR, TAR and TBR).

CONTACTS AND LOCATIONS:
Overall Officials: Yogish Kudva, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials